CLINICAL TRIAL: NCT00272363
Title: Clinical and Molecular Studies in Families With Glaucoma and Related Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060059; 06-EI-0059
Record Dates: First submitted 2006-01-05; First posted 2006-01-05 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2016-07-29

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective

SUMMARY:
This study will document the clinical and genetic features of glaucoma and related diseases, including normal tension glaucoma (NTG). Researchers would like to define genetic influences and eventually isolate the genes causing those diseases.

Glaucoma is an important cause of vision loss in the United States and worldwide. The disease is marked by a wearing down of the retina and optic nerve, often associated with increased pressure in the eye. It is often an inherited trait. This study will involve between 250 and 2,000 patients over a 5-year period. It will examine the natural history of the genotype, or genetic makeup, of a person and the phenotype, that is, visible situations produced by the interaction of the genotype and one's environment.

Patients 4 and older who have glaucoma or related diseases or whose family members have those diseases may be eligible for this study. They will complete a medical history for the doctors to verify the diagnosis, inquire about medical problems and surgical operations, and gather data about vision problems in a patient's family (by drawing a family tree). The complete eye examination may take several hours. Eye drops will be used to dilate, or enlarge, the pupils of patients' eyes, and the pupils will stay dilated for 4 to 6 hours. There may be some temporary glare in brightly lit areas, which can be reduced by wearing of sunglasses. Patients may experience some blurring of vision. There may be a localized allergic reaction to the medication used or an increase of pressure inside the eye. If that occurs, medication to control the reaction will be given. In addition, photographs of the retina and perhaps even the lens will be taken. For that procedure, eye drops will dilate the pupils of the eyes. The light that is involved with the specialized photography may cause some mild discomfort. Patients will undergo eye tests regarding color vision, field of vision, and ability to see the dark. Also, there will be a measurement of pressure in the eye and thickness of the cornea.

To study patients' DNA, the researchers will obtain a blood sample of about 4 teaspoons from patients 10 years or older. A smaller amount of about 1 teaspoon for each 5 lb. of body weight will be collected from younger patients. Those DNA samples will be used only for research in the genetic disorder in a patient's family. No other testing or research will be conducted on the blood samples without patients' separate permission. Also, the DNA will be stored by codes that the researchers define and contained in a secured building.

In this study, researchers will not provide information about a patient's health to patient family members or to other people. They will not discuss information such as adoption or biological fatherhood unless it has medical implications for the patient or the patient's family members.

If information obtained from this study may be important to patients' health, they will be informed when it is available. There are no plans to give patients the results of any medical tests, evaluations, or other research data. Further research may be needed before such results become meaningful.

DETAILED DESCRIPTION:
Objective: This project, Clinical and Molecular Studies in Families with Glaucoma and Related Diseases, will study the inheritance of glaucoma in families of many nationalities and ethnic backgrounds in order to identify the genes that, when mutated, cause glaucoma, elevated intraocular pressure, or similar diseases and the pathophysiology through which they act.

Study Population: The number of subjects to be enrolled has no logical upper limit, but will be at least 250 and not more than 2000 during the next 5 years.

Design: The study consists of ascertaining individuals and especially families with multiple individuals, affected by glaucoma or related retinal and anterior chamber diseases. These patients and their families will undergo detailed ophthalmological examinations and, where indicated, additional non-investigational examinations to characterize disease in their families and determine their affectation status. A blood sample will be collected from each individual for isolation of DNA and in some individuals biochemical testing or for lymphoblastoid transformation to establish a renewable source of DNA. Linkage analysis, physical mapping, SNP and microsatellite analysis for association studies, and mutational screening will be carried out to identify the specific the gene and the mutations in it that are associated with glaucoma in this family. If necessary, the gene product or blood sample will be characterized biochemically. The study will enroll subjects at the NEI and at collaborating institutions.

Outcome Measures: Linkage will be determined using the lod score method and mutations in specific genes will be assessed using a combination of residue conservation, blosum score, and molecular modeling. Biochemical, metabolic, and physiological effects will be individualized to the specific assay.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects with the following will be recruited:

1. Individuals or family members of individuals with glaucoma, either congenital, childhood, or age related.
2. Adults must be capable of providing their own consent.
3. All subjects must be able to cooperate with study examination and phlebotomy.
4. Older than 4 years of age.

EXCLUSION CRITERIA:

1. Diseases, infections, or trauma that mimic primary glaucoma.
2. Children requiring sedation for study procedures.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2005-12-29; Study Completion 2016-07-29

PRIMARY OUTCOMES:
Statistically significant linkage | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: James F Hejtmancik, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (4):
- United States (3):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Duke University, Durham, North Carolina
  - University of Utah, Salt Lake City, Utah
- Eye Research Institute, Zhongstan Ophthalmic Ctr, Sun Yat-Sen University, Guangzhou, China

REFERENCES:
- [Background] Kubota R, Kudoh J, Mashima Y, Asakawa S, Minoshima S, Hejtmancik JF, Oguchi Y, Shimizu N. Genomic organization of the human myocilin gene (MYOC) responsible for primary open angle glaucoma (GLC1A). Biochem Biophys Res Commun. 1998 Jan 14;242(2):396-400. doi: 10.1006/bbrc.1997.7972. PMID 9446806
- [Background] Leske MC, Nemesure B, He Q, Wu SY, Fielding Hejtmancik J, Hennis A. Patterns of open-angle glaucoma in the Barbados Family Study. Ophthalmology. 2001 Jun;108(6):1015-22. doi: 10.1016/s0161-6420(01)00566-8. PMID 11382622
- [Background] Nemesure B, He Q, Mendell N, Wu SY, Hejtmancik JF, Hennis A, Leske MC; Barbados Family Study Group. Inheritance of open-angle glaucoma in the Barbados family study. Am J Med Genet. 2001 Sep 15;103(1):36-43. doi: 10.1002/ajmg.1498. PMID 11562932